CLINICAL TRIAL: NCT00792649
Title: Comparison Between HD+ Endoscopy and Standard Videoendoscopy in Screening Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Hoffman Arthur, Hoffman Arthur
Other Study IDs: 837.386.07
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-02

CONDITIONS: Polyps; Neoplasia
MeSH Terms: conditions — Polyps; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: screening colonoscopy with HD+ endoscopes
- 2: screening colonoscopy with standardvideoendoscopes

SUMMARY:
Colonoscopy is the accepted gold standard for screening of colorectal cancer. However, small and flat neoplastic lesions might be overlooked with standard video endoscopes. The new available EPKi system (Pentax, Japan) enables with HD+ imaging resolution above HDTV standard. Aim of the study was to test the efficacy of HD+ colonoscopy alone and in conjunction with I-Scan (newly developed post processing digital filter)in comparison to standard videoendoscopy

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients scheduled for screening colonoscopy

Exclusion Criteria:

* Inflammatory bowel disease
* Cancer
* Pregnancy
* Inability to obtain informed consent
* Prothrombin time < 50% of control
* Partial thromboplastin time > 50 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients scheduled for screening colonoscopy were examined using HD+ colonosccopes and standardendoscopes.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-02